CLINICAL TRIAL: NCT04373161
Title: Utilizing Home Pulse Oximetry for Patients With COVID-19 To Monitor Disease Progression
Brief Title: Home Pulse Oximeter Use in Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Hospital (Other)
Responsible Party: Principal Investigator, Kaushal Majmudar, Physician, Swedish Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020032301
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Sars-CoV2; COVID-19; COVID
Keywords: Oximetry; Oximeter; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Suspected COVID-19 patients being discharged to home (Experimental): Patients will be given a portable, fingertip pulse oximeter to take home. Patients will monitor their resting home oxygen saturation three times per day.
  Interventions: Device: Home Pulse Oximetry Monitoring

INTERVENTIONS:
Device: Home Pulse Oximetry Monitoring — Patients to check their home oxygen saturation three times daily and return to the ED for sustain oxygen <92% or for worsening symptoms.

SUMMARY:
The purpose of this study is to investigate the use of home pulse oximetry monitoring in patients with COVID-19 to trend disease progression and identify need for hospitalization.

DETAILED DESCRIPTION:
This protocol studies patients with suspected non-severe Corona Virus Disease (COVID-19) being discharged to home from an emergency department (ED) or outpatient testing center. Patients will be provided a portable fingertip home pulse oximeter that measures peripheral oxygen saturation (SpO2). Patients will be instructed to check their resting home oxygen saturation three times per day and record these findings. They will be instructed to return to the emergency room for sustained oxygen saturation below 92% or if their symptoms are worsening and they feel they need medical attention. Patients will be called once daily by the research team to collect data in real time. Patients will be monitored for seven days, and at the end of the seven day period, they will return the pulse oximeter as well as a spreadsheet of their home oximetry readings. The purpose is to see if home pulse oximetry identifies disease progression and need for hospitalization in patients with COVID-19. Additionally, there will be analysis of trends in home oximetry readings wand predictors of morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected COVID-19 as defined by the World Health Organization
* Age > 18

Exclusion Criteria:

* Pregnancy
* Prisoners
* Lack of decision making capacity or cannot provide consent
* Patients being admitted to the hospital
* Patients on home oxygen
* Patients being discharged to a skilled nursing facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
Hospitalization in COVID-19 patients with low home SpO2 | 7 days after enrollment
  The primary outcome is the relative risk of hospitalization in COVID-19 patients with resting home pulse oximeter SpO2 below 92%.

SECONDARY OUTCOMES:
Trend in resting home pulse oximetry readings | 7 days after enrollment
  The purpose of this outcome is to determine if home pulse oximetry readings abruptly drop, gradually decline, or stay level in patients with COVID-19
Timing of SpO2 <92% | 7 days after enrollment
  This will evaluate if there is a correlation between the time of day with SpO2 readings below 92 percent in patients with suspected COVID-19.
Home pulse oximeter use effect on subsequent ED visits | 7 days after enrollment
  The goal of this outcome is to see if patients enrolled in the study are reassured by use of home pulse oximeter monitoring and if this device prevents subsequent ED visits by patients
Reason for return to the Emergency Department | 7 days after enrollment
  To see if patients who return to the ED and end up hospitalized did so for incidental finding of low home pulse oximetry or if it was for worsening symptoms
Hospitalization outcome - morbidity | Up to 21 days after enrollment
  The study will assess development of morbidity defined as intensive care unit admission, acute respiratory distress syndrome, and/or septic shock in patients with SpO2 <92%
Hospitalization outcome - mortality | Up to 21 days after enrollment
  The study will assess mortality defined as death after admission to the hospital in patients with SpO2 <92%
Median Length of Stay | Up to 21 days after enrollment
  The study will measure median length of stay in patients with COVID-19 that are hospitalized on subsequent return to the ED.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Shah, DO, Study Director — Swedish Hospital
Locations (1):
- Swedish Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No